CLINICAL TRIAL: NCT04854148
Title: Validation of a Smartphone-based Assessment of Movement Health Compared to a Battery of Standardized Clinical Tests for Mobility, Stability, and Posture
Brief Title: Validation of a Smartphone-based Assessment of Movement Health
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Shirley Ryan AbilityLab (Other)
Responsible Party: Principal Investigator, Arun Jayaraman, PT, PhD, Principle Investigator, Shirley Ryan AbilityLab
Other Study IDs: STU00214468
Record Dates: First submitted 2021-04-16; First posted 2021-04-22 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2022-05

CONDITIONS: Mobility Limitation
MeSH Terms: conditions — Mobility Limitation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Experimental: Each participant will perform a Smartphone movement health assessment and a series of 12 gold standard tests under the supervision of a licensed physical therapist or other research study staff
  Interventions: Other: Smartphone Movement Health Assessment

INTERVENTIONS:
Other: Smartphone Movement Health Assessment — Participants will perform the assessment using an App installed on a smartphone device. Following the smartphone assessment, gold standard clinical assessments will be performed and scored for comparison
  Other Names: Gold Standard Movement Assessments

SUMMARY:
To correlate a smartphone-based assessment of mobility, stability, and posture with those derived from standard clinical tests among a heterogeneous cohort.

DETAILED DESCRIPTION:
Smartphone movement health assessment introduces a new measure of health that helps users analyze and improve their mobility, stability and posture through performance of movements and physical exercises. To verify the accuracy of this measure, the goal is to provide data-driven evidence regarding its accuracy in comparison to gold standard tests for measuring movement health. To address this challenge, the assessment scores will be benchmarked to a set of gold standard tests and sensor metrics for measuring movement health recommended by professional associations such as the American Physical Therapy Association (APTA) or American College of Sport Medicine (ACSM) and found valid in clinical studies , .

ELIGIBILITY:
Inclusion Criteria:

1. All participants should be able to perform the Smartphone movement health assessment and receive a score for their movement health. This will be evaluated by the research team members during the recruitment process.
2. Ages 18-85 years old
3. Able and willing to give written consent and comply with study procedures

Exclusion Criteria:

1. Pregnant or nursing
2. Skin allergies or irritation that would prevent safe use of sensors described in protocol

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Community-dwelling adults
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2021-04-21 (Actual); Primary Completion 2022-12-12 (Estimated); Study Completion 2022-12-12 (Estimated)

PRIMARY OUTCOMES:
Correlation | Baseline
  Positive correlation between Smartphone's movement health assessment scores and the scores of standardized tests and sensors metrics for mobility, stability and posture

CONTACTS AND LOCATIONS:
Overall Officials: Arun Jayaraman, PT, PhD, Principal Investigator — Shirley Ryan AbilityLab
Locations (1):
- Shirley Ryan AbilityLab, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided